CLINICAL TRIAL: NCT03593733
Title: Comparison Between Photobiomodulation Therapy (PBMT) and a Cold-Water Immersion (CWI) in Recovery Soccer Player: Analysis of Biochemical Markers of Recovery and Muscular Oxidative Stress.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: LUCIANA MARIA MALOSA SAMPAIO (Other)
Responsible Party: Sponsor-Investigator, LUCIANA MARIA MALOSA SAMPAIO, Professor of Postgraduate Program in Rehabilitation Science, University of Nove de Julho
Organization: University of Nove de Julho (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PBTM CWI
Record Dates: First submitted 2018-06-25; First posted 2018-07-20 (Actual); Last update posted 2024-05-07 (Actual); Status verified 2024-05

CONDITIONS: Soccer; Fatigue; Oxidative Stress; Recovery; Cold Water Immersion; Photobiomodulation Therapy
MeSH Terms: conditions — Fatigue | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold Water Immersion (Experimental): Cold Water Immersion
  Interventions: Other: Cold Water Immersion
- Photobiomodulation Therapy (Experimental): Photobiomodulation Therapy
  Interventions: Other: Photobiomodulation Therapy

INTERVENTIONS:
Other: Photobiomodulation Therapy — Photobiomodulation Therapy
  Other Names: Cold Water Immersion
  Arms: Photobiomodulation Therapy
Other: Cold Water Immersion — Cold Water Immersion
  Arms: Cold Water Immersion

SUMMARY:
Competitive soccer engages many of the body's systems to a major extent. The musculoskeletal, nervous, immune and metabolic systems are stressed to a point where recovery strategies post-exercise become influential in preparing for the next match.

Recovery from exercise can be an important factor in performance during repeated bouts of exercise. In a tournament situation, where athletes may compete numerous times over a few days, enhancing recovery may provide a competitive advantage. Recent work has highlighted that the aim of most recovery interventions is to return psychological, physiological, and performance variables to the 'pre-exercise' level or to baseline conditions identified in the absence of fatigue.

The post-exercise cold water immersion (CWI) through its primary ability to decrease tissue temperature and blood flow, is purported to facilitate recovery by ameliorating hyperthermia and subsequent alterations to the central nervous system (CNS), reducing cardiovascular strain, removing accumulated muscle metabolic by-products, attenuating exercise-induced muscle damage (EIMD) and improving autonomic nervous system function. All these alterations provoke important physiological changes for the recovery of the athlete.

Scientific evidence for other strategies reviewed in their ability to accelerate the return to the initial level of performance is still lacking. These include active recovery, stretching, compression garments, massage and electrical stimulation. While this does not mean that these strategies do not aid the recovery process, the protocols implemented up until now do not significantly accelerate the return to initial levels of performance in comparison with a control condition.

Among these new strategies, Photobimodulation therapy - PBMT using low-level laser therapy (LLLT) and light-emitting diode therapy (LEDT) has been the focus of important research insights science in recent years. The PBMT has been used to increase muscle performance and reduces muscle fatigue signals. The mechanism proposed for the use of PBMT in sports and exercise is the increase in cytochrome c-oxidase in skeletal muscle fibers that lead to upregulation of mitochondrial activity, which increases ATP production promoting more energy for the muscle and decreases oxidative stress and reactive oxygen species production.

Considering that the consented CWI is already used with good results in soccer athletes, however it has some drawbacks such as the time of application and the inconvenience caused by the application of cold and the new possibilities presented in the literature of the use of PBMT we propose to carry out this study. To address these issues, the present study aims to investigate and analyze biological markers on oxidative stress and muscle damage in soccer athletes after a match submitted to recovery strategies through CWI and PBMT

DETAILED DESCRIPTION:
In elite soccer, players are frequently required to play consecutive matches interspersed by 3 days and complete physical performance recovery may not be achieved. Incomplete recovery might result in underperformance and injury. During congested schedules, recovery strategies are therefore required to alleviate post-match fatigue, regain performance faster and reduce the risk of injury. Recovery from exercise can be an important factor in performance during repeated bouts of exercise.

The strenuous exercise induces muscle cell structural damage, which results in increased plasma concentrations of muscle enzymes such as CK and LDH. The efflux of CK and LDH proteins from muscle may be attributed to increased permeability of the plasma membrane or intramuscular vasculature (or both). Thus, a reduction in these markers has been proposed as an indicator of recovery after strenuous exercise that induces muscle damage.

ELIGIBILITY:
Inclusion Criteria:Voluntary athletes were soccer players aged 16 to 17 years, healthy, male, with no history of autoimmune diseases, who did not present previous muscular lesions in the period of 3 months prior to the study and who are participating of the category championships.

-

Exclusion Criteria:

* No soccer playres.

Ages: 16 Years to 17 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Serum levels of Creatine Kinase (CK) activity | Baseline; immediatily soccer match and 48 hours after.
  Sample of Blood
Serum levels Thiobarbituric acid reactive substances -TBARS | Baseline; immediatily soccer match and 48 hours after.
  Sample of Blood
Serum levels Superoxide Dismutase -SOD | Baseline; immediatily soccer match and 48 hours after.
  Sample of Blood
Serum levels Catalase - CAT | Baseline; immediatily soccer match and 48 hours after.
  Sample of Blood

CONTACTS AND LOCATIONS:
Overall Officials: Paulo de Tarso Camillo de Carvalho, Professor, Principal Investigator — University of Nove de Julho

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Versey NG, Halson SL, Dawson BT. Water immersion recovery for athletes: effect on exercise performance and practical recommendations. Sports Med. 2013 Nov;43(11):1101-30. doi: 10.1007/s40279-013-0063-8. PMID 23743793
- [Background] Ihsan M, Watson G, Abbiss CR. What are the Physiological Mechanisms for Post-Exercise Cold Water Immersion in the Recovery from Prolonged Endurance and Intermittent Exercise? Sports Med. 2016 Aug;46(8):1095-109. doi: 10.1007/s40279-016-0483-3. PMID 26888646
- [Background] Nedelec M, McCall A, Carling C, Legall F, Berthoin S, Dupont G. Recovery in soccer : part ii-recovery strategies. Sports Med. 2013 Jan;43(1):9-22. doi: 10.1007/s40279-012-0002-0. PMID 23315753
- [Background] Vanin AA, Verhagen E, Barboza SD, Costa LOP, Leal-Junior ECP. Photobiomodulation therapy for the improvement of muscular performance and reduction of muscular fatigue associated with exercise in healthy people: a systematic review and meta-analysis. Lasers Med Sci. 2018 Jan;33(1):181-214. doi: 10.1007/s10103-017-2368-6. Epub 2017 Oct 31. PMID 29090398
- [Background] de Oliveira AR, Vanin AA, Tomazoni SS, Miranda EF, Albuquerque-Pontes GM, De Marchi T, Dos Santos Grandinetti V, de Paiva PRV, Imperatori TBG, de Carvalho PTC, Bjordal JM, Leal-Junior ECP. Pre-Exercise Infrared Photobiomodulation Therapy (810 nm) in Skeletal Muscle Performance and Postexercise Recovery in Humans: What Is the Optimal Power Output? Photomed Laser Surg. 2017 Nov;35(11):595-603. doi: 10.1089/pho.2017.4343. PMID 29099680
- [Background] De Marchi T, Schmitt VM, Machado GP, de Sene JS, de Col CD, Tairova O, Salvador M, Leal-Junior EC. Does photobiomodulation therapy is better than cryotherapy in muscle recovery after a high-intensity exercise? A randomized, double-blind, placebo-controlled clinical trial. Lasers Med Sci. 2017 Feb;32(2):429-437. doi: 10.1007/s10103-016-2139-9. Epub 2017 Jan 5. PMID 28054262
- [Result] Reilly T, Ekblom B. The use of recovery methods post-exercise. J Sports Sci. 2005 Jun;23(6):619-27. doi: 10.1080/02640410400021302. PMID 16195010
- [Result] Nedelec M, McCall A, Carling C, Legall F, Berthoin S, Dupont G. Recovery in soccer: part I - post-match fatigue and time course of recovery. Sports Med. 2012 Dec 1;42(12):997-1015. doi: 10.2165/11635270-000000000-00000. PMID 23046224
- [Result] Wilcock IM, Cronin JB, Hing WA. Physiological response to water immersion: a method for sport recovery? Sports Med. 2006;36(9):747-65. doi: 10.2165/00007256-200636090-00003. PMID 16937951
- [Result] Murray A, Cardinale M. Cold applications for recovery in adolescent athletes: a systematic review and meta analysis. Extrem Physiol Med. 2015 Oct 12;4:17. doi: 10.1186/s13728-015-0035-8. eCollection 2015. PMID 26464795